CLINICAL TRIAL: NCT05415969
Title: Uremic Pruritus Among Adults on Dialysis in the French Speaking Part of Switzerland
Brief Title: CKD-aP Among Adults on Dialysis in Switzerland
Acronym: UP-RAISE
Status: Completed | Type: Observational
Sponsor: University of Applied Sciences of Western Switzerland (Other)
Collaborators: University of Lausanne Hospitals (Other); Hôpital Fribourgeois (Other); University Hospital, Geneva (Other); Valais Hospital (Unknown); eHnv Hospital (Unknown); Rennaz Hospital (Unknown); Intercantonal Hospital of Broye (Unknown); GHOL Nyon Hospital (Unknown); Dialyse Riviera (Unknown); Cecil Clinic Hirslanden Private Hospital Group (Unknown); Vifor Pharma (Industry); Réseau Hospitalier Neuchâtelois (Other)
Responsible Party: Principal Investigator, Nancy Helou, Full Professor UAS, University of Applied Sciences of Western Switzerland
Other Study IDs: 2022-00670
Record Dates: First submitted 2022-06-01; First posted 2022-06-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Kidney Diseases; Dialysis; Chronic Kidney Diseases Associated Pruritus
Keywords: Chronic Kidney Disease; Dialysis; Pruritus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CKD-aP — Identification of CKD-aP prevalence and severity among patients on dialysis.

SUMMARY:
Chronic Kidney Disease Associated Pruritus (CKD-aP) represents a localized or a generalized skin itch, which is a common symptom occurring in end-stage renal disease and dialysis. The prevalence of CKD-aP in adults on dialysis varies between countries ranging between 20-42%. Swiss data on CKD-aP are unfortunately largely lacking, as Switzerland is so far not part of large registries, such as DOPPS.

The aging population, the increase in diabetes (69% by 2030), the increase in hypertension (60% by 2025) and poly-morbidity will probably lead to a rise in the number of patients on dialysis and subsequent CKD-aP.

CKD-aP is associated with sleep disturbances, compromised quality of life, emotional distress, and increased risks of hospitalization and death. Its management lacks approaches that are supported by strong evidence because its pathogenesis remains poorly understood and may be related to an increase in uremic toxins, skin inflammation. In this context, sweat composition deserves more attention.

Aim of the study The aim of the study is to determine the prevalence of CKD-aP in the population on dialysis, the association between CKD-aP and different electrolytes, and the potential role of the composition of sweat in CKD-aP.

Results will be used for building a CKD-aP symptom management program to improve the quality of care of patients on dialysis and will be incorporated in the nursing continuing education program.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years old
* Diagnosed with end-stage renal disease and receiving hemodialysis for at least 6 months
* Able to communicate in French or availability of a French-speaking close relative for translation
* Signed informed consent

Additional inclusion criteria for the case-control study outcomes phase 2:

* Reporting moderate to severe CKD-aP for the participant considered as a case
* Reporting no or mild CKD-aP for the participant considered as a control Cases and controls will be matched by age-group, sex, and dialysis modality (hemodialysis or peritoneal dialysis).

Exclusion Criteria:

* Presence of cognitive impairment or cognitive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients on hemodialysis or peritoneal dialysis followed by nephrologists in private and public hospitals of the French speaking Part of Switzerland.
Sampling Method: Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of CKD-aP | June 27, 2022- October 31, 2023
  Evaluation of the presence of CKD-aP. This outcome prevalence will be reported in %.
Severity of CKD-aP using the Visual Analog Scale | June 27, 2022- October 31, 2023
  Severity of CKD-aP will be measured using the Visual Analog Scale (VAS) questionnaire. Participants will be asked to rate their maximum pruritus intensity during the last 24 hours.
  The VAS score ranges from 0 (not itchy) to 10 (extremely itchy); Severity will be classified into five categories: 1) 0 = no pruritus, 2) 0.1-2.9 points = mild pruritus, 3) 3.0-6.9 points = moderate pruritus, 4) 7.0-8.9 points = severe pruritus, and 5) 9.0-10.0 points = very severe pruritus. Higher scores indicate a worse outcome.
Severity of CKD-aP using the Verbal Rating Scale | June 27, 2022- October 31, 2023
  Severity of CKD-aP will also be measured using the Verbal Rating Scale (VRS) questionnaire. Participants will be asked to rate their maximum pruritus intensity during the last 24 hours.
  The VRS is a five-point scale and consists of a list of adjectives describing various levels of symptom intensity (0= no itch, 1= mild itch, 2= moderate itch, 3= severe itch and 4=very severe itch). Higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Sodium level (mmol/l) in sweat | June 27, 2022- October 31, 2023
  Measurement of sodium (mmol/l) in a subgroup of patients with CKD-aP and their age-sex-matched controls on dialysis.
  60 participants (30 cases and 30 controls)
Chloride level (mmol/l) in sweat | June 27, 2022- October 31, 2023
  Measurement of chloride (mmol/l) in a subgroup of patients with CKD-aP and their age-sex-matched controls on dialysis.
  60 participants (30 cases and 30 controls)
Potassium level (mmol/l) in sweat | June 27, 2022- October 31, 2023
  Measurement of potassium (mmol/l) in a subgroup of patients with CKD-aP and their age-sex-matched controls on dialysis.
  60 participants (30 cases and 30 controls)
Calcium level (mg/l) in sweat | June 27, 2022- October 31, 2023
  Measurement of calcium (mg/l) in a subgroup of patients with CKD-aP and their age-sex-matched controls on dialysis.
  60 participants (30 cases and 30 controls)
Phosphorus level (mg/ml) in sweat | June 27, 2022- October 31, 2023
  Measurement of phosphorus (mg/ml) in a subgroup of patients with CKD-aP and their age-sex-matched controls on dialysis.
  60 participants (30 cases and 30 controls)
Urea level (mmol/l) in sweat | June 27, 2022- October 31, 2023
  Measurement of urea (mmol/l) in a subgroup of patients with CKD-aP and their age-sex-matched controls on dialysis.
  60 participants (30 cases and 30 controls)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized Data can be shared upon justified request.